CLINICAL TRIAL: NCT01565733
Title: Multicenter, Open Label, Non-randomized, Non-interventional Observational Study of Safety of Treatment Initiation With a Biphasic Insulin Aspart (NovoMix® 30) in Hospitalized Patients With Type 2 Diabetes Mellitus
Brief Title: Safety of Treatment Initiation With Biphasic Insulin Aspart 30 in Hospitalised Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-4017
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovoMix® 30 users
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Biphasic insulin aspart 30 prescribed solely on the basis of clinical judgement. Initial dose, frequency of injections and further dosage amendments at the discretion of the treating physician.

SUMMARY:
This study is conducted in Europe. The aim of this study is to evaluate the safety and efficacy of biphasic insulin aspart (NovoMix® 30) in hospitalised patients with type 2 diabetes with the aim of intensifying their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Treated with oral anti-diabetics and/or human insulin

Exclusion Criteria:

* Persons previously included in the trial
* Hypersensitive to biphasic insulin aspart or any of the excipients
* Pregnant or lactating women, or those who plan to get pregnant within the next 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes requiring treatment with NovoMix® 30 insulin on admission who before hospitalisation had been treated with oral antidiabetics and/or human insulin
Sampling Method: Non-Probability Sample
Enrollment: 2223 (Actual)
Dates: Start 2007-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Frequency of severe hypoglycaemic episodes

SECONDARY OUTCOMES:
Number of severe hypoglycaemic episodes
Number of mild hypoglycaemic episodes
Postprandial glucose concentration after breakfast, lunch, and dinner
Average fasting glucose concentration after waking and before main meals
Average plasma glucose level at bedtime and at night

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Warsaw, Poland

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com